CLINICAL TRIAL: NCT07285317
Title: Ensayo Exploratorio Para Evaluar la Tolerancia de Una Bacteria Con Potencial probiótico (Phascolarcobacterium Faecium) de Nueva generación Para Proteger la Salud metabólica en Humanos
Brief Title: Safety and Tolerability Evaluationof Phascolarcobacterium Faecium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spanish National Research Council (Other Government)
Responsible Party: Principal Investigator, Yolanda Sanz Herranz, Professor, Spanish National Research Council
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 217/2023
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Health; Obesity Type 2 Diabetes Mellitus; Obesity & Overweight
Keywords: Gut microbiota; Obesity; Metabolic health; Probiotic; Phascolarctobacterium faecium
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: This study uses a parallel interventional model with two predefined groups: normal-weight individuals and individuals with overweight and mild alterations in glucose metabolism. All participants receive Phascolarctobacterium faecium. All participants follow the same intervention and assessment schedule, allowing for within-group comparisons before and after supplementation, as well as exploratory analyses between the two population subgroups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P. faecium in healthy normal weight individuals (Experimental): Healthy normal weight individuals will receive a daily dose of P. faecium for 15 days to evaluate the tolerability and safety of short-term administration.
  Interventions: Dietary Supplement: Bacterium P. faecium
- P. faecium in overweight individuals with mild alterations in glucose homeostasis (Experimental): Overweight individuals with mild alterations in glucose homeostasis will receive P. faecium for 15 days to evaluate its safety and tolerability in the target population.
  Interventions: Dietary Supplement: Bacterium P. faecium

INTERVENTIONS:
Dietary Supplement: Bacterium P. faecium — The participants will be given Phascolarctobacterium faecium orally (pill form) for 15 consecutive days.

SUMMARY:
The goal of this interventional study is to assess the safety and tolerability of the daily administratrion of bacterium Phascolarctobacterium faecium in healthy adults with normal weight, and in individuals with overweight and alterations in glucose metabolism. The main questions this study aims to answer are:

Is the bacterium intake safe? Is the bacterium intake well tolerated? The objecitves are to assess if the intake of the bacterium is well tolerated by assessing gastrointenstinal symptoms, and safe, by assessing biochemical markers, incidence of adverse events and the general health status.

Participants will take daily the bacterium for 15 days. Study assessments include stool collection for microbiota analysis; blood sampling form biochemical tests, anthropometric measurements, and validated questionnaires on diet, physical activity, and perceived health.

DETAILED DESCRIPTION:
A total of 20 adult volunteers will consume a daily dose of Phascolarctobacterium faecium once per day for 15 consecutive days. Stool and blood samples will be collected at baseline and after the intervention; blood draws will be performed following an overnight fasting of at least 8 hours. Participants will also complete online questionnaires assessing sociodemographic characteristics, gastrointestinal symptoms, bowel habits, general health status, physical activity, and dietary habits. In addition, body composition parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* stable body weight and dietary habits during the previous three months
* written informed consent

Exclusion Criteria:

* the presence of gastrointestinal disorders
* immunodeficiency
* eating disorders
* antibiotic use within one month before the study
* chronic antidiabetic therapy
* substance (drug) abuse
* restrictive diets
* any other condition deemed inappropriate for participation by the clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and general health status | 21 days
  Participants will have access to a 24-hour contact number to report any inconvenience or adverse effects. All adverse effects will be recorded throughout the intervention period and for one additional week after completion. Outcomes will be reported as the presence or absence of adverse effects.
Systemic safety of P. faecium intake assessed in all the clinical trial participants by biochemical markers | 15 days
  Complete hemogram and biochemical analysis will be permormed at baseline and after bacterum intervention and includes red blood cells, white blood cells, and assessments of lipid profile (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol, and non-HDL cholesterol), renal function (urea, creatinine, and uric acid), hepatic function (total protein, AST, and ALT), and glucose homeostasis (glucose, insulin, HbA1c, and HOMA-IR).
  All parameters will be measured using standard units commonly applied in clinical practice, and results will be compared before and after the intervention. It will be interpreted as either unchanged or altered relative to baseline values.
Tolerability assessment measured by stool habit | 15 days
  To assess the tolerability of P. faecium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, capturing both weekly bowel movement frequency and stool consistency using the Bristol Stool Scale. Stool habits will be evaluated by integrating these two variables: a normal habit will be defined as 4-14 bowel movements per week together with a Bristol score of 3-5, whereas any deviation from these ranges will be classified as an altered stool habit.
Tolerability assessment measured by the frequency of heartburn. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of heartburn. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.
Tolerability assessment measured by the frequency of abdominal bloating. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of abdominal bloating. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.
Tolerability assessment measured by the frequency of constipation. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of constipation. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.
Tolerability assessment measured by the frequency of diarrhea. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of diarrhea. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.
Tolerability assessment measured by the frequency of nausea. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of nausea. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.
Tolerability assessment measured by the frequency of flatulence. | 15 days
  Use of probiotic bacteria may occasionally elicit mild gastrointestinal discomfort, including bloating, gas or abdominal cramps. To assess the tolerability of the tested bacterium, participants will complete gastrointestinal symptom questionnaires before and after the intervention, which also capture the frequency of flatulence. Response options include: "all the time," "most of the time," "sometimes," "a few times," and "never." Changes in frequency will be compared between pre- and post-treatment assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Sanz, Professor, Principal Investigator — Instituto de Agroquímica y Tecnología de Alimentos (IATA-CSIC)
Locations (1):
- Instituto de Agroquímica y Tecnología de Alimentos (IATA-CSIC), Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Xu Z, Zhang J. A comparison of nursing education curriculum in China and the United States. J Nurs Educ. 2002 Jul;41(7):310-6. doi: 10.3928/0148-4834-20020701-07. No abstract available. PMID 12137122